CLINICAL TRIAL: NCT01002144
Title: C-Reactive Protein as a Predictor for Airway Hyper-responsiveness
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: the sponsor is the principal investigator, Rambam Health Care Campus
Other Study IDs: CRPAHR - CTIL
Record Dates: First submitted 2009-09-30; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood sampling

SUMMARY:
Background: Increased serum high sensitivity C-reactive protein (hs-CRP) has been associated with airway inflammation in asthma and may serve as a surrogate marker for the presence of airway hyper-responsiveness (AHR) in this set-up. This study was designed to evaluate the predictive value of hs-CRP for AHR assessed by metacholine challenge test (MCT), in adults with suspected Asthma.

ELIGIBILITY:
Inclusion Criteria:

* subjects that were referred to Metacholine challenge test

Exclusion Criteria:

* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people with suspected asthma underwent metacholine chalange test.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Yigla, MD, Principal Investigator — Rambam Health Care Campus